CLINICAL TRIAL: NCT04433819
Title: Skin Microcirculation Evaluation With Nailfold Capillaroscopy in Cushing's Syndrome Patients
Brief Title: Nailfold Capillaroscopy Evaluation in Cushing Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.474
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cushing Syndrome; Hypercortisolism
Keywords: Cushing's syndrome; Capillaroscopy; Cushing's disease; Adrenal adenoma; Nailfold capillary; Microvascular circulation
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cushing syndrome: Male and female patients diagnosed as Cushing syndrome caused by ACTH-producing pituitary adenoma or cortisol producing adrenal adenoma
- Controls: Healthy controls matched for age, gender, and body mass index

SUMMARY:
This cross-sectional, single-center study will assess the microvascular function using a nailfold video-capillaroscopy in patients with endogenous Cushing syndrome.

DETAILED DESCRIPTION:
Endogenous Cushing's syndrome (CS) is associated with increased macrovascular diseases and impaired endothelial function. There is no clear data about the effects of hypercortisolism on microcirculation.

The primary aim of this study is to evaluate the peripheric microvascular area in patients with Cushing's syndrome. The association of microvascular changes with present comorbidities (diabetes, hypertension, etc.) and disease activation will be evaluated.

Method:

Cushing syndrome patients admitted to our clinic will be included in this study for the next six months after given informed consent.

The following clinical laboratory parameters will be evaluated as cross-sectionally.

Previous medical history, available laboratory parameters (fasting plasma glucose, HbA1c, total cholesterol, triglyceride, HDL, LDL, creatine, AST, ALT, complete blood count, ACTH, dexamethasone suppression tests (1 mg- 2mg), urine free cortisol, FSH, LH, total testosterone, estradiol, IGF-1, TSH, free T3, free T4, prolactin), radiologic images (Cranial MRI and Adrenal MRI) will be recorded from medical charts.

Nailfold microcirculation will be evaluated with video-capillaroscopy: it is a non-invasive atraumatic assessment of the morphology and some functional aspects of cutaneous capillaries.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed as Cushing syndrome (CS) caused by ACTH-producing pituitary adenoma or cortisol producing adrenal adenoma
* Age between 18 and 70 years

Exclusion Criteria:

* Chronic glucocorticoid use
* CS caused by ectopic ACTH producing tumors
* CS caused by adrenocortical carcinoma
* Pseudo CS
* Patients with Raynaud phenomenon
* Patients with collagen tissue disease
* Patients who use drugs that affect the metabolism of fibrinolysis (such as oral contraceptives)
* Employees at work at risk of microtrauma (such as gardeners, farmers)
* Skin diseases with nail fold involvement (such as dermatitis, psoriasis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed as endogenous Cushing syndrome, and age and sex matched controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Nailfold capillary number of tortuous loops | 6 months
  Nailfold capillary area changes
Nailfold capillary area number of meandering capillaries | 6 months
  Nailfold capillary area changes
Nailfold capillary avascular areas | 6 months
  Nailfold capillary area changes

SECONDARY OUTCOMES:
Correlation between nailfold capillary number of tortuous loops and presence of diabetes | 6 months
  Independent risk factors that affected nailfold capillaroscopy images
Correlation between nailfold capillary number of tortuous loop with urine free cortisol levels | 6 months
  Presence and severity of hypercortisolism as an independent risk factor

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Gogas Yavuz, M.D., Study Director — Marmara University School of Medicine, Endocrinology and Metabolism Department
Locations (1):
- Marmara University Medical School Section of Endocrinology and Metabolism, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No